CLINICAL TRIAL: NCT04149600
Title: Identification of Genetic Causes of Calcific Aortic Valve Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Simon Robson, Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2018P000380
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Calcific Aortic Stenosis; Calcific Aortic Stenosis - Bicuspid Valve; Aortic Valve Disease; Aortic Valve Calcification; Aortic Diseases; Aortic Aneurysm; Aortic Valve Cusp Abnormality; Aortic Valve Disease Mixed; Aortic Valve Insufficiency
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Disease; Aortic Diseases; Aortic Aneurysm; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Broadly, in order to perform the study, we will collect DNA for genotyping and "discarded" aortic valve and aortic tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bicuspid aortic valve: We wish to investigate the etiology of calcific aortic valve disease, and aortic dilation or aneurysm in patients with a bicuspid aortic valve undergoing aortic valve replacement or aortic surgery.
  Interventions: Procedure: Patients scheduled to undergo aortic valve replacement or aortic surgery at BIDMC will be approached for participation in this study.
- Tricuspid aortic valve: Data and samples will be compared using a control group comprised of patients with a tricuspid aortic valve undergoing aortic surgery.
  Interventions: Procedure: Patients scheduled to undergo aortic valve replacement or aortic surgery at BIDMC will be approached for participation in this study.

INTERVENTIONS:
Procedure: Patients scheduled to undergo aortic valve replacement or aortic surgery at BIDMC will be approached for participation in this study. — Adult patients undergoing aortic valve replacement (AVR) and/or aortic resection will be enrolled.

SUMMARY:
This study aims to identify the molecular genetic causes of the variability in development of calcific aortic valve disease in bicuspid and tricuspid aortic valves and their associated aortic dilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a plan to undergo elective aortic valve replacement and/or ascending aortic surgery

Exclusion Criteria:

* Age < 20 years
* Unable/unwilling to consent
* History of aortic valve replacement or transcatheter aortic valve replacement (TAVR)
* History of endocarditis
* History of rheumatic fever
* History of chest radiotherapy
* History of organ transplant

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators wish to identify the molecular genetic causes of the variability in development of calcific aortic valve disease and aortic dilation in patients with a plan to undergo elective aortic valve replacement and/or ascending aortic surgery at BIDMC.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of expression signatures of aortic valve development and calcification in the macroscopically normal and abnormal portions of aortic valves excised during aortic valve replacement. | 8 years
  We will take a portion of the aortic valve and/or aortic tissue that is routinely excised for aortic valve or aortic replacement for expression analyses and generation of fibroblast cell lines. In collaboration with the Department of Pathology, we have established methods to take sufficient "normal" and abnormal tissue while allowing formal routine pathological evaluation.
  All tissue samples for expression analysis will be transported in iced RNALater and later frozen in a -80°C research freezer, prior to next generation sequencing. We may use tissue samples to develop cell lines for indefinite use.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No